CLINICAL TRIAL: NCT03439644
Title: Physiological Upper Eyelid Laxity
Acronym: LAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: LAX
Record Dates: First submitted 2018-02-08; First posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Eyelid Laxity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurement of the upper eyelid laxity — Measurement using a soft slider of the distance between our 2 marks The difference obtained between the measurement and the initial 10 millimeters corresponds to the tarsal laxity.

SUMMARY:
This is a prospective, single-center study in normal subjects aged 20 to 89 years.

The objective was to describe upper eyelid laxity by age group (20/29 years old, 30/39 years old, 40/49 years old, 50/59 years old, 60/69 years old, 70/79 years old and 80/89 years old) measured with the method of McNab and studying it according to her customary side of sleep. In addition, we evaluated a method for measuring tarsal laxity.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 89 years
* be free
* be able to give informed consent

Exclusion Criteria:

* History of facial paralysis, upper palpebral trauma or palpebral surgery
* History of sleep apnea syndrome
* Impossibility to give consent
* Pregnant or lactating women
* Persons enjoying enhanced protection and persons deprived of their liberty by a judicial or administrative decision

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Evolution of upper eyelid laxity | 10 minutes
  Comparison of upper right and left palpebral laxity values in millimeters between different age groups

CONTACTS AND LOCATIONS:
Overall Officials: Roxane FLAUSSE, Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU DE Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided